CLINICAL TRIAL: NCT01402648
Title: Effects of the Dietary Supplementation With a Blend of ER Beta Agonists on the Expression of ER Beta and Related Biomarkers of Cell Proliferation and Apoptosis, in Sporadic Colon Adenopolyposis
Brief Title: Estrogen Receptor Beta Agonists (Eviendep) and Polyp Recurrence
Acronym: CRC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CM&D Pharma Limited (Industry)
Responsible Party: Alfredo Di Leo, Head Gastroenterology Unit, D.E.T.O. - University Hospital, Bari (Italy)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CMD-CRC09(2)
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Adenocarcinoma of Colon Recurrent
Keywords: Non adenomatous mucosa; Estrogen Receptor beta and apoptosis; Adenoma recurrence; Screening colonoscopy every 3-5 years; patients at intermediate risk for CRC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary supplement (Placebo Comparator): 900 mg Maltodextrins
  Interventions: Dietary Supplement: Maltodextrins
- Eviendep (CM&D Pharma Limited, UK) (Active Comparator): 175 mg milk thistle (fruit dry extract, 70% in silymarin)+ 20 mg flaxseed (dry extract, 40% in secoisolariciresinoldiglucoside) + 750 mg non starch, insoluble and indigestible fiber (6% in lignin).
  Interventions: Dietary Supplement: Eviendep (CM&D Pharma Limited, UK)

INTERVENTIONS:
Dietary Supplement: Eviendep (CM&D Pharma Limited, UK) — 175 mg milk thistle (fruit dry extract, 70% in silymarin)+ 20 mg flaxseed (dry extract, 40% in secoisolariciresinoldiglucoside)+750 mg non-starch, insoluble and indigestible fiber (6% in lignin). Provided in 5 g sachets, to be dissolved in half glass water, administered twice a day for 60 days on top of the common diet.
  Arms: Eviendep (CM&D Pharma Limited, UK)
Dietary Supplement: Maltodextrins — 900 mg maltodextrin+excipient as per the active comparator eviendep, up to 5 g/sachet
  Arms: Dietary supplement

SUMMARY:
The decreased Estrogen Receptor beta (ERβ) expression in the non adenomatous mucosa of ApcMin/+ mice favours intestinal neoproliferation. The dietary supplementation with a blend of ERβ agonists and lignin has been shown to recover ERβ to the healthy wild type levels, and a reduced polyp number and lower dysplasia was also observed in the adenomatous mucosa. In this randomised, double blind and placebo controlled study, we assessed if ERβ similarly guides the apoptotic control of cell proliferation in the non adenomatous colon mucosa of patients affected from sporadic adenopolyposis, prone to polyp recurrence. For 60 day in advance of the screening colonoscopy, patients were supplemented with a dietary blend of ERβ agonists and lignin (Eviendep, CM&D Pharma Limited, London, UK) on top their common diet (left unchanged during the study period), to study if the pro-proliferative behavior of the non adenomatous mucosa was effected. Sixty patients naïve from previous and concomitant hormonal or anti-inflammatory CRC chemoprevention were sequentially 1:1 randomised to active or placebo supplementation. ERα and ERβ (mRNA, Western Blotting, Elisa, immunostaining), TUNEL, caspase-3 and Ki-67 (immunostaining) were assessed in bioptic normal colon mucosa samples. Study power: 80%, type 1 error: .05 (two-tails). Statistics: Non parametric Wilcoxon test for efficacy. MANOVA for proliferative and apoptotic biomarkers relationships to the common diet and to the 60 day supplementation.

DETAILED DESCRIPTION:
Enrolled patients were actively ongoing the surveillance program for the follow up of polyp recurrence and progression to CRC. Eligible patients should have undergone a polypectomy since 2003, affected by multiple polyps < 10 mm or one-two adenomas < 10 mm and/or with a grade of dysplasia to make them classified at intermediate risk for CRC, and scheduled to screening colonoscopy each 3-5 years. Patients were sequentially 1:1 randomly allocated to placebo or Eviendep at baseline (T0). The dietary supplements were administered twice a day for 60 days in advance of the screening colonoscopy, thus covering approximately eight complete colon epithelial turnover to occur. Five days in advance of T60 colonoscopy, patients refrained from fresh and cooked fruit and vegetable intake. Bowel cleansing was achieved by PEG 4000 oral administration (1120 g/4 L water solution). N=8 biopsy samples/patient were collected from the non adenomatous mucosa in the sigmoidal colon. Small polyps (diameter less or equal 0.5 cm) were topically electrocoagulated, whereas villous and tubulovillous polyps (diameter equal or higher than 0.5 cm) were submitted to the histological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age: 50-70 years
* Menopausal women since at least 2 years
* Diagnosed since 2003 for adenomas, underwent polypectomy and histological assessment
* Regularly inscribed and actively ongoing the surveillance program for the follow-up of adenoma recurrence and progression to advanced adenomas
* Screening colonoscopy every 3-5 years
* No previous or concomitant administration of ASA and NSAIDs
* No previous or concomitant administration of Hormonal Replacement Therapy (HRT)
* No previous or concomitant administration of other phytoestrogens

Exclusion Criteria:

* Chronic inflammatory intestinal disease
* Intestinal and/or extraintestinal malignant neoplasms
* Acute or chronic renal disease
* Anemia
* Coagulation disorders,
* BMI > 30
* Systemic corticosteroids
* Anticoagulants or platelet antiaggregants
* Antibiotics within 30 days from enrollment

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Expression of ERβ, ERα, TUNEL, Caspase-3, Ki-67 in bioptic samples of non adenomatous mucosa in sporadic adenopolyposis | 60 days following dietary oral supplementation, in advance of the screening colonoscopy as per the planning of the surveillance program
  ERβ and ERα protein content (Elisa), mRNA and immunohistochemically stained cells (% over the total number of cells/field,ICH); TUNEL (%,ICH); caspase-3 (%,ICH), Ki-67 (%ICH), and comparison (mean, median, %ICH) between study groups. Safety assessed by no induction of ERα expression.

SECONDARY OUTCOMES:
Safety assessed by unchanged hematochemistry | 30 and 60 days following dietary oral supplementation
  Hemoglobin ≥ 12.0 g/dL; platelets ≥ 120,000/mm3; INR ≤ 1.5; AST or ALT ≤ 1.5 times the upper limit of normal values (ULN); Alkaline Phosphatase ≤ 1.5 times ULN; Bilirubin ≤ 1.5 times ULN; BUN ≤ 40 mg/dL; normal blood pressure or controlled hypertension
Urinary lignans | baseline (T0, 30 (T30) and 60 (T60) days during the study period
  To verify comparability of phytoestrogens contributed from the common diet in the two arms at baseline, and to assess compliance to the active comparator during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Policlinico Consorziale - Gastroenterology Unit, Bari, Bari, Italy